CLINICAL TRIAL: NCT06345131
Title: Clinical Research Plan for the Safety and Accuracy of Ultrasound-guided Radial Artery
Brief Title: Clinical Research Plan for the Safety and Accuracy of Ultrasound-guided Radial Artery Puncture Catheterization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Liu Han, associate professor, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20230829-06
Record Dates: First submitted 2024-01-30; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Surgical Patients
Keywords: Ultrasound guidance; Radial artery

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transverse diameter of radial artery (TDA) (Other): The patient was placed in a supine position, the upper limb was abducted on the operative side, the palm was upward, and the wrist joint was extended at an angle of 45°.Radial artery puncture catheterization is performed within this group
  Interventions: Other: Non invasive blood pressure monitoring
- vertical distance of radial artery (center) from skin (VDA) (Other): The patient was placed in a supine position, the upper limb was abducted on the operative side, the palm was upward, and the wrist joint was extended at an angle of 45°.Radial artery puncture catheterization is performed within this group
  Interventions: Other: Non invasive blood pressure monitoring
- distance of superficial branch of radial nerve relative to horizontal position of radial artery (D) (Other): The patient was placed in a supine position, the upper limb was abducted on the operative side, the palm was upward, and the wrist joint was extended at an angle of 45°.Radial artery puncture catheterization is performed within this group
  Interventions: Other: Non invasive blood pressure monitoring

INTERVENTIONS:
Other: Non invasive blood pressure monitoring — Non invasive blood pressure monitoring

SUMMARY:
By observing the anatomical relationship and influencing factors of the radial artery through ultrasound, the optimal puncture location is selected, and puncture catheterization is guided to reduce the number of punctures, reduce complications, and improve safety and accuracy.

DETAILED DESCRIPTION:
Measure the anatomical parameters of the radial artery and radial nerve in the forearm using ultrasound, summarize the relevant anatomical factors that affect the placement of radial artery catheterization, and find the optimal puncture range that is both safe and accurate for radial artery catheterization.

A total of 100 surgical patients were included. Ultrasound was used to measure the transverse diameter (TDA) of the radial artery, the vertical distance (VDA) between the radial artery (center) and the skin, and the distance (D) between the superficial branch of the radial nerve and the radial artery at the midpoint between the radial styloid process point, 2.5cm, 5cm, 7.5cm, 10cm from the radial styloid process point, 2.5cm below the center of the elbow fossa, and 10cm from the radial styloid process point and 2.5cm below the center of the elbow fossa. The radial artery was compared on both sides of the patient, as well as on different genders and ages Differences in anatomical parameters and spatial relationships of the radial nerve. Patients were randomly divided into a distal group (Group A, 33 cases), a mid distal group (Group B, 33 cases), and a proximal group (Group C, 33 cases). Group A underwent radial artery puncture and catheterization within 0-5cm of the proximal end of the radial styloid process; Group B underwent radial artery puncture and catheterization within 5-10cm of the proximal end of the radial styloid process; Group C underwent radial artery puncture and catheterization within a range of 10cm proximal to the styloid process of the radius and 2.5cm below the center of the cubital fossa. The success rate, puncture time, puncture frequency, and puncture related complications of the first ultrasound-guided radial artery puncture and catheterization were recorded for three groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Selected surgical patients planning to undergo general anesthesia and invasive arterial blood pressure monitoring
2. ASA grading I to II
3. Age 18-65
4. Agree to participate in this clinical study and sign an informed consent form

Exclusion Criteria:

1. Patients with positive or suspected positive Allen test
2. Peripheral vascular diseases
3. Coronary artery related diseases
4. Local skin infections, ulcers, scars, and surgical history
5. Shock patients or receiving cardiac stimulants, vasoconstrictors, etc
6. Peripheral nerve injury, anatomical abnormalities, and neurological dysfunction
7. Passive upper limb position, unable to cooperate in completing ultrasound assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Measure the transverse diameter of the radial artery at each anatomical point | Before anesthesia surgery
  The patient is in a flat lying position, with both upper limbs abduction, palms facing upwards, and wrist joint angle of 45 °. A portable ultrasound instrument (probe frequency 13-6MHz, Sono Sound Company) is used, and the ultrasound probe is in vertical contact with the forearm in the short axis direction, Explore the relative anatomical sites of the radial artery (confirmed by Doppler) on the left and right sides of the body surface projection line of the radial artery (from 2.5cm below the center of the cubital fossa to the inner side of the radial styloid process), with a relative distance of 2cm. There is no significant compression of the radial artery during scanning to maintain the normal shape and location of the blood vessels.

CONTACTS AND LOCATIONS:
Overall Officials: Han Liu, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutwein A, Thalhammer C. Ultrasound-guided venous pressure measurement. Vasa. 2022 Nov;51(6):333-340. doi: 10.1024/0301-1526/a001032. Epub 2022 Oct 6. PMID 36200379
- [Background] Genre Grandpierre R, Bobbia X, Muller L, Markarian T, Occean BV, Pommet S, Roger C, Lefrant JY, de la Coussaye JE, Claret PG. Ultrasound guidance in difficult radial artery puncture for blood gas analysis: A prospective, randomized controlled trial. PLoS One. 2019 Mar 20;14(3):e0213683. doi: 10.1371/journal.pone.0213683. eCollection 2019. PMID 30893349
- [Background] Maitra S, Baidya DK, Ray BR, Chowhan G, Bhattacharjee S. Comparison of ultrasound guided dorsal radial artery cannulation and conventional radial artery cannulation at the volar aspect of wrist: A pilot randomized controlled trial. J Vasc Access. 2023 Nov;24(6):1463-1468. doi: 10.1177/11297298221093953. Epub 2022 Apr 26. PMID 35470717

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-07-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT06345131/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-07-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT06345131/SAP_001.pdf